CLINICAL TRIAL: NCT01271296
Title: Use of Liquorice and Grapefruit in Patients With Addison's Disease
Brief Title: Effects and Interactions of Liquorice and Grapefruit on Glucocorticoid Replacement Therapy in Addison's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Lars Birger Nesje, Head of Department of Medicine, Haukeland University Hospital, Helse-Bergen HF, Haukeland University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 3.2007.2620 (REK); 17775 (NSD) (Other: Norwegian Social Science Data Services (registry for approval of data protection)); 07/5829 (SHdir) (Other: The Norwegian Directorate of Health and Social Affairs (Approval of research biobank)); 3.2007.2620 (Other: West Regional Committee of Research Ethics)
Record Dates: First submitted 2010-12-22; First posted 2011-01-06 (Estimated); Last update posted 2011-01-17 (Estimated); Status verified 2010-12

CONDITIONS: Addison Disease
Keywords: Addison Disease; Pharmacokinetics; Hormone Replacement Therapy; cortisone acetate; Quality of Life
MeSH Terms: conditions — Addison Disease | interventions — Glycyrrhiza glabra extract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Liquorice (Active Comparator): Liquorice eq to 150 mg glycyrrhizinic acid. Results are compared to a baseline assessment without liquorice/grapefruit juice ingestion.
  Interventions: Dietary Supplement: Liquorice
- Grapefruit juice (Active Comparator): 200 ml pink grapefruit juice three times a day. Results are compared to a baseline assessment without liquorice/grapefruit juice ingestion.
  Interventions: Dietary Supplement: Grapefruit Juice
- Baseline (No Intervention): Baseline assessment without intake of liquorice or grapefruit juice

INTERVENTIONS:
Dietary Supplement: Liquorice — 24 gram liquorice eq. to 150 mg glycyrrhizinic acid, taken orally, for three days.
  Arms: Liquorice
Dietary Supplement: Grapefruit Juice — 200 ml pink grapefruit juice three times a day, taken orally, for three days.
  Arms: Grapefruit juice

SUMMARY:
Addison's disease is a rare disease, wherein the adrenals can not produce sufficient steroid hormones (cortisol and aldosterone). Patients with Addison's disease report impaired subjective health status, and they have increased all-cause mortality. Conventional therapy is by oral replacement of glucocorticoid and mineralocorticoid hormones, but this strategy imperfectly mimic the diurnal cortisol variations, and render the patients both over- and under-treated. Anecdotally, some patients with adrenal insufficiency may benefit from the use of various nutritional compounds. We hypothesised that liquorice and grapefruit altered the metabolism and absorption of cortisone acetate.

DETAILED DESCRIPTION:
In the present study, cortisone acetate absorption and metabolism are assessed in subjects with Addison's disease on three occasions. On the first occasion, the subjects are on their regular diet, but avoid ingestion of grapefruit and liquorice. At the end of the baseline assessment the order of the nutritional compounds (liquorice-grapefruit juice or grapefruit juice-liquorice) to be investigated in the next two assessments are randomised.

On the two next occasions, the absorption and metabolism of cortisone acetate is studied when study subjects consume liquorice and grapefruit juice. Between the use of grapefruit and liquorice there is a wash out period of at least 3 weeks.

For studies on liquorice effects, the subjects ingest 24-gram liquorice per day (equivalent of 150-mg glycyrrhizinic acid per day). For studies on grapefruit juice effects, subjects drink 200-ml grapefruit juice three times a day for three days. They maintain their regular medication and usual diet.

Time-series of cortisol and cortisone are obtained in serum and saliva samples on the third day of liquorice/grapefruit juice use. 24-hour urine is also collected.

Measurements of cortisol and metabolites in serum and saliva are used to calculate pharmacokinetical parameters. The measurements from samples obtained when using the investigated nutritional compounds are compared to the baseline assessment in each subject. Metabolites in 24-hour urine are compared similarly to investigate changes in urinary excretion, and to estimate the activity of enzymes involved in the metabolism of cortisol (5alfa-reductase, 5beta-reductase, cytochrome P450 3A4 system, 11-beta hydroxysteroid dehydrogenase).

ELIGIBILITY:
Inclusion Criteria:

* Verified diagnosis of adrenal insufficiency (Addison's disease)
* Stable cortisone acetate replacement therapy
* Written informed consent

Exclusion Criteria:

* Malignant disease
* Pharmacological treatment with other glucocorticoids
* Pregnancy
* Current minor disease (ie the flu)
* Major disease or accident requiring hospitalization the last three months
* Use of grapefruit juice or liquorice the last two weeks before study start
* Blood pressure above 150mmHg systolic or 90 mmHg diastolic.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
AUC Serum Cortisol - Levels of cortisol in serum during the first 2.6 hours after oral administration of cortisone acetate. | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  The area under the curve (AUC) of cortisol is calculated based on serum time-series sampling (every 20 minutes for 2.6 h after oral administration of cortisone acetate). The AUCs obtained during liquorice and grapefruit juice intakes are compared to the baseline assessment (without these nutritional compounds). All other pharmacokinetic properties (primary and secondary outcome measures) are compared analogously.

SECONDARY OUTCOMES:
Serum Cortisol levels at the end of time-series sampling (t=160min) | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  At the end of time series sampling (160 minutes after orally administered cortisone acetate) on all three assessments
Serum Cortisone levels at the end of time-series sampling (t=160min) | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  At the end of time series sampling (160 minutes after orally administered cortisone acetate) on all three assessments
Saliva Cortisol levels at the end of time-series sampling (t=160min) | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  At the end of time series sampling (160 minutes after orally administered cortisone acetate) on all three assessments
Saliva Cortisone levels at the end of time-series sampling (t=160min) | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  At the end of time series sampling (160 minutes after orally administered cortisone acetate) on all three assessments
Time of maximum concentration of serum Cortisol | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  Based on time-series sampling at each of the three assessments
Time of maximum concentration of serum Cortisone | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  Based on time-series sampling at each of the three assessments
Time of maximum concentration of Saliva Cortisol | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  Based on time-series sampling at each of the three assessments
Time of maximum concentration of Saliva Cortisone | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  Based on time-series sampling at each of the three assessments
Half life of serum cortisol | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  Based on time-series sampling at each of the three assessments
Half life of serum cortisone | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  Based on time-series sampling at each of the three assessments
Urinary aTHF/THF-ratio | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  Measured in 24h urine obtained at the three assessments.
  aTHF = allo-tetrahydrocortisol, THF = tetrahydrocortisol
AUC Serum Cortisone | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  Similar to primary outcome Serum AUC Cortisol
Urine total metabolites (Urinary cortisol+cortisone+6OHF+aTHF+THF+THE) | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  24-hour urine collected on each of the three assessments
  aTHF = allo-tetrahydrocortisol, THF = tetrahydrocortisol, THE = tetrahydrocortisone, 6OHF = 6beta-hydroxycortisol
Urinary ratio (aTHF+THF)/THE | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  Assessed in 24h urine obtained at the three assessments (baseline, after liquorice and after grapefruit juice). It is an index of 5-reductase activity.
  24-hour urine collected on each of the three assessments
  aTHF = allo-tetrahydrocortisol, THF = tetrahydrocortisol, THE = tetrahydrocortisone
Urinary Ratio Cortisol/6beta-OH-Cortisol | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  Assess the enzymatic activity of CYP3A4 by the index urinary cortisol/6beta-oh cortisol ratio obtained at the three assessments (baseline, after liquorice and after grapefruit juice.
  6OHF = 6beta-hydroxycortisol
Urine total metabolites (Urinary cortisol+cortisone+6OHF+aTHF+THF+THE) | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  24-hour urine collected on each of the three assessments
  24-hour urine collected on each of the three assessments
  aTHF = allo-tetrahydrocortisol, THF = tetrahydrocortisol, THE = tetrahydrocortisone, 6OHF = 6beta-hydroxycortisol
AUC Saliva cortisone | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  Similar to primary outcome Saliva AUC Cortisol, but for cortisone.
AUC Serum Cortisone | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  Similar to primary outcome Serum AUC Cortisol, but for cortisone.
AUC Saliva Cortisol | Outcome measures are assessed when all subjects have completed the study, approximately 1.5-2.0 years after study start.
  Similar to AUC Serum Cortisol, but measurements are on saliva.

CONTACTS AND LOCATIONS:
Overall Officials: Paal Methlie, MD, Principal Investigator — University of Bergen. Helse-Bergen HF; Kristian Løvås, MD, PhD, Principal Investigator — University of Bergen. Helse-Bergen HF.; Eystein S Husebye, Prof, MD, Principal Investigator — University of Bergen. Helse-Bergen HF.; Ernst A Lien, Prof. MD., Principal Investigator — University of Bergen
Locations (1):
- Haukeland University Hospital, Helse-Bergen HF, Bergen, Norway